CLINICAL TRIAL: NCT01956071
Title: Workers' Acceptability of a Prototype Integrated and Interactive Pedal Desk
Acronym: WAPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principle Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PBRC 2013-050
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-10

CONDITIONS: Acceptability of Semi-recumbent Pedal Desk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WAPD (Experimental): Participants were asked to complete three tasks while simultaneously pedaling at a sustainable and self-selected pace. The three tasks were: 1) compose and send an email; 2) search a topic on the internet, and 3) complete an on-line questionnaire.
  Interventions: Device: WAPD

INTERVENTIONS:
Device: WAPD — The objective was to assess workers' acceptability of the Pennington Pedal Desk.

SUMMARY:
The purpose of this study is to assess full-time workers'impressions and acceptability of a prototype pedal desk. The pedal-desk is a semi-recumbent (upright) portable pedal mechanism that allows workers to complete tasks in a traditional seated position.

DETAILED DESCRIPTION:
Researchers in recent years have begun to consider how modern occupational practices and environments could be enriched to facilitate increased energy expenditure by replacing sedentary behaviors with opportunities for non-exercise physical activity without competing with time committed to work tasks. The investigators have developed a pedal desk: a semi-recumbent (upright) portable pedal mechanism with a maneuverable and adaptable desktop. While utilizing the pedal desk, workers are able to complete their tasks in a more traditional seated position. Determining workers' acceptability is a key initial step in translating this "sedentary behavior countermeasure" to real workplace settings.

In addition to having their height, weight, body fat percentage, and bioelectrical impedance measured, eligible participants will be asked to complete three tasks while simultaneously pedaling at a sustainable and self-selected pace. The three tasks are: 1) compose and send an email; 2) search a topic on the internet, and 3) complete an on-line questionnaire. The questionnaire that participants will complete was developed specifically for this study, utilizes Likert scales, and is based on the Theory of Planned Behavior. Constructs tested focus on perceptions of using the pedal desk at work and include: behavioral beliefs, normative beliefs, control beliefs, intention, self-efficacy, and an open-ended question soliciting general impressions concerning using the pedal desk at work.

ELIGIBILITY:
Inclusion Criteria:

* full-time employee at Pennington Biomedical Research Center
* between ages 21 and 65
* self-report primarily sitting while at work
* comfortable sending emails and searching topics on the internet

Exclusion Criteria:

* weigh more than 250 pounds
* have physical limitations that prevent performance of pedaling motions
* pregnancy
* pacemaker or metal joint replacement

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Full time employees of Pennington Biomedical Research Center will be invited by email to participate in an on-line screening survey. The on-line survey will include a series of questions to determine eligibility.
Groups:
- Pedal Desk Acceptability: Orientation sessions will last approximately 30 minutes and will provide participants detailed information about the study, including the number and type of assessments, the length and nature of the pedal desk trial session, the time commitment required, and the potential risks and benefits of participation. Participants will be given a copy of the informed consent form to read and review. Interested participants will schedule their 30 minute trial visit.
  At the trial visit, participants' questions will be answered and they will be asked to complete the informed consent form prior to beginning any study procedures. At this one and only visit height, weight, body fat percentage, and Bioelectrical Impedance Analysis will be measured. Participants will also be asked to complete 3 computer based tasks while using the pedal desk (1) search a topic on the internet; (2) compose and send an email, and (3) complete an on-line questionnaire while utilizing the pedal desk.
Period: Overall Study
Arm/Group | Pedal Desk Acceptability
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pedal Desk Acceptability
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Pedal Desk Trial Questionnaire
Description: Full-time sedentary workers used the pedal desk for 15 minutes while they: 1) searched the internet, 2) composed an email, and 3) completed acceptability ratings using an online Likert scale anchored from 1/strongly disagree to 5/strongly agree. The Questionnaire assessed subjective opinions about exercise and use of the Pedal Desk. No subscale or total scores were generated, and there are no maximum or minimum values. Rather, the number and proportion of participants who rated "strongly agree", etc. on each item was calculated.
Time Frame: Visit 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pedal Desk Acceptability
Number analyzed (Participants) | 42
Participants
  Agree: can complete usual tasks while pedaling | 41
  Disagree: can complete usual tasks while pedaling | 1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Pedal Desk Acceptability
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes